CLINICAL TRIAL: NCT03164031
Title: A Clinical Trial Evaluating the Feasibility and Acceptability of Orthotic Shorts for Walking Function in People With Multiple Sclerosis.
Brief Title: Feasibility and Acceptability of Orthotic Shorts for People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2016-7/HWB-HSC-14
Record Dates: First submitted 2017-04-11; First posted 2017-05-23 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be trialling two different pairs of shorts, where one pair will be designed as an orthoses and the other will look similar but be looser and not designed to support the hips.
  The investigator is also the main outcome assessor and they will be blinded to which pair of shorts will be worn at each stage of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Close-fitting orthotic shorts condition (Experimental): Orthotic shorts will be made to measure for each participant, designed to provide some compression to the hips, pelvis and thighs and to provide support. Shorts will be worn during objective testing of walking ability and then taken home. Wear will be increased gradually over 5 days but then worn every day during normal daily activity.
  Interventions: Device: Close-fitting orthotic shorts
- Looser fitting shorts condition (Active Comparator): Looser shorts will be made to measure for each participant, designed to look similar to the orthotic shorts but provide minimal support or compression. Shorts will be worn during objective testing of walking ability and then taken home. Wear will be increased gradually over 5 days but then worn every day during normal daily activity.
  Interventions: Device: Looser fitting shorts

INTERVENTIONS:
Device: Close-fitting orthotic shorts — The orthotic shorts will be custom-made by DM Orthotics, a UK based company that specialises in dynamic, elastomeric orthoses for healthcare and sport. They will provide both pairs of shorts for each participant, both constructed from a 275 g/m2 fabric, which is 51% Polyamide, 32% Dorlastan and 17% cotton. A company representative will assess each participant to decide the compression and fit of the shorts, such as whether support for the lower trunk is required. The shorts can be manufactured with a toileting hole, if preferred, allowing participants to toilet without removing the shorts. Shorts with a toileting hole are worn beneath usual underwear.
  Other Names: Lycra garment, Dynamic Elastomeric Fabric Orthosis
  Arms: Close-fitting orthotic shorts condition
Device: Looser fitting shorts — Looser fitting shorts will be custom-made by DM Orthotics, a UK based company that specialises in dynamic, elastomeric orthoses for healthcare and sport. Shorts will be constructed from a 275 g/m2 fabric, which is 51% Polyamide, 32% Dorlastan and 17% cotton. A company representative will assess each participant to decide the fit of the shorts. The shorts can be manufactured with a toileting hole, if preferred, allowing participants to toilet without removing the shorts. Shorts with a toileting hole are worn beneath usual underwear.
  Arms: Looser fitting shorts condition

SUMMARY:
Walking can be slow and unsteady in people with multiple sclerosis (MS). This study will investigate whether orthotic shorts might help.

Orthotic shorts are similar to the tight clothing believed to improve performance in athletes. Research suggests that such shorts help stroke survivors to walk faster. Some people with MS find that similar garments improve coordination and stability. Public funding is controversial because there is no research investigating whether they work in people with MS.

This is a cross-over study in which participants will each trial two different pairs of shorts. The first aim is to determine whether these shorts are acceptable to people with MS. Secondly, the study will develop the tools required to test the shorts. For example, by determining which measures seem most appropriate and if specific factors predict whether the shorts might help. The hypothesis being tested is that the shorts are acceptable.

People with MS will be invited to participate in this mixed methods study, aiming for a sample size of 16 people. Participants will trial two different pairs of shorts, one of which will fit more closely than the other. The shorts will be tested in a movement laboratory and in daily life.

In the movement laboratory, participants will be measured in both pairs of shorts and in normal, loose clothing. Walking pattern, speed and variability will be measured when the shorts are first worn.

Participants will test shorts in their normal daily life for up to two weeks. They will complete questionnaires about their walking and balance in the different shorts and record how long they wear the shorts. Interviews will explore expectations and experiences of the shorts and of the research study.

In the analyses, data from interviews will be combined with the numerical information gained from laboratory measures, diaries and questionnaires. If the shorts are acceptable, this study will inform a larger trial investigating effectiveness.

DETAILED DESCRIPTION:
Study design - This is a mixed methods, randomised cross-over study investigating two different pairs of orthotic shorts. The shorts will be tested in two main ways, firstly, the impact of the shorts on objectively assessed walking ability when first worn and, secondly, acceptability and impact of the shorts on self-perceived ability over a two-week period when the shorts are worn in the community.

Participants - Participants will be people with multiple sclerosis (PwMS) who identify themselves as having some difficulty walking, with a lack of stability around the hips and/or lower trunk. The study aims to recruit 16 PwMS over a 15-16-month period. It is felt that a sample size of 16 will enable the shorts to be trialled with participants with a range of different movement problems as well as different ages, genders and activity levels. These characteristics may impact upon the effect and acceptability of the shorts.

Recruitment - Participants will be made aware of the study through flyers, online advertisements and in discussion with local healthcare professionals. Potential participants will be identified through a local neurological therapy service.

Procedure - Each participant will visit Sheffield Hallam University on four occasions and be seen at home on three occasions.

The first Sheffield Hallam visit (Appointment 1) will include informed consent, collection of basic participant details, an initial interview around expectations and motivations, completion of self-report measures, assessment and measurement for shorts with a representative from the orthotics company and provision of a falls diary for completion over the following two weeks. Participants will be randomly assigned to the order in which the different shorts will be tested.

The second and third Sheffield Hallam visits (Appointments 3 and 5) follow the same structure with each visit testing one of the two pairs of shorts. Firstly, walking ability without the shorts will be measured. They will put the shorts on and spend about 30 minutes becoming familiar with wearing the shorts before the objective measures are repeated. After the objective assessments, participants will be provided with further information on wearing and caring for the shorts and a wear diary and falls diary to be completed whilst the shorts are trialed at home.

The final Sheffield Hallam visit (Appointment 7) will include a final measure of walking ability without shorts plus a semi-structured interview around the participants' experiences of the shorts and the trial.

In between the above visits to Sheffield Hallam, there will be three shorter visits. Each participant can choose to attend university or meet in an agreed location if preferred. The first of these (Appointment 2) will be with the representative from the orthotics company to check the fit of the shorts and measure the pressure exerted by the shorts. If adjustments are required at this point, this will be done within 3 days and the shorts will then be delivered to the chief investigator. Appointments 4 and 6 are to collect the shorts, the diaries and the self-report measures reporting the perceived impact of the shorts after the period of home wear.

Intervention - The orthotic shorts will be custom-made by a UK based company that specialises in dynamic, elastomeric orthoses for healthcare and sport. They will provide two pairs of shorts for each participant, which will differ in the closeness of their fit. The company representative, who will assess each participant, will decide the compression and fit of the shorts, such as whether support for the lower trunk is required. The shorts can be manufactured with a toileting hole, if preferred, allowing participants to toilet without removing the shorts. Shorts with a toileting hole are usually worn beneath usual underwear.

Randomisation and allocation - Counter-balancing will ensure that half the group use the more closely fitting shorts first and half the looser shorts first. A randomisation schedule will be created by a using the Sealed Envelope online system for blocked randomisation. Shorts will be placed into sealed envelopes labelled "Shorts 1" and "Shorts 2" by a third party using the randomisation schedule.

Data collection - Semi-structured interviews will be conducted on two occasions for each participant - at the first appointment and at the final appointment.

At Appointment 1, participants will be interviewed to explore their motivations for joining the study, their expectations of the shorts, their current daily activities and their readiness for change. The data from this interview will enable investigation of whether certain aims, motivations or perceptions impact upon the eventual acceptability of the shorts. This initial interview is likely to last 20 - 40 minutes.

At Appointment 7, participants will be interviewed about their experiences during the study. This interview aims to determine the acceptability of the shorts and participants' views on the study processes such as the information and support they received, and the outcome measures used. Prior to the interview, the interviewer will review the data and reflective notes from the initial interview; the wear diaries and the Participant Global Rating of Change scores at the initial assessment and will use this information to inform the questions that are asked. This will ensure the interviews are focussed on aspects that are important to each participant. This final interview is likely to last 40 - 60 minutes.

Measures of walking ability - Outcome measures are described elsewhere and have been chosen according to current guidelines on the most relevant assessment battery for walking in PwMS. In addition to movement laboratory measures, participants will complete self-report assessments of their walking and balance; a falls diary and a rating of the overall impact on the shorts on their walking ability.

Data analysis - Qualitative and quantitative data will first be analysed separately and then combined, partly by transforming qualitative into categorical data where this provides a valid representation of the data and partly by comparing, contrasting and relating the findings of the different data types for each objective.

Qualitative data analysis will use the Framework Approach to thematic analysis.

Descriptive quantitative data analysis will determine individual and average changes on each measure and effect sizes for the impact of the shorts. Effect sizes will indicate which measures are most responsive to this intervention and this information may be used to inform a sample size calculation for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having multiple sclerosis of any type (relapsing-remitting, primary progressive or secondary progressive).
* Clinically stable - have not experienced relapse in the last 4 weeks; have not commenced a novel therapy in the last 3 months.
* Able to travel to Sheffield Hallam University for assessments.
* Have difficulty walking with a subjective feeling of instability around the hips or lower trunk.
* Able to walk for at least 2 minutes at a time.
* Able to provide a written record of informed consent.

Exclusion Criteria:

* People who do not meet inclusion criteria.
* Skin conditions that may be exacerbated by tight clothing.
* Circulatory problems that may be exacerbated by tight clothing, such as varicose veins, previous thrombosis, venous or arterial insufficiency.
* Cognitive problems including memory disturbance that may impact on recall of experience and adherence to guidance.
* Pregnancy - because of related circulatory problems.
* Living further than 10 miles from Sheffield if they are unable to provide own transport and the home visits would be too far for the researcher to travel.
* Have previously used orthotic shorts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Adherence to wear protocol | After two weeks of shorts wear
  Adherence will be calculated as hours worn as a percentage of hours of wear requested.

SECONDARY OUTCOMES:
Cadence | At baseline and on Day 1 of shorts wear
  A GAITRite system will be used to assess spatio-temporal gait parameters. Participants will walk 4 times over a 5.18m walkway.
Step length | At baseline and on Day 1 of shorts wear
  A GAITRite system will be used to assess spatio-temporal gait parameters. Participants will walk 4 times over a 5.18m walkway.
Proportion of gait cycle in double support | At baseline and on Day 1 of shorts wear
  A GAITRite system will be used to assess spatio-temporal gait parameters. Participants will walk 4 times over a 5.18m walkway.
Width of base of support | At baseline and on Day 1 of shorts wear
  A GAITRite system will be used to assess spatio-temporal gait parameters. Participants will walk 4 times over a 5.18m walkway.
Variability of step length | At baseline and on Day 1 of shorts wear
  A GAITRite system will be used to assess spatio-temporal gait parameters. Participants will walk 4 times over a 5.18m walkway.
Variability of stride time | At baseline and on Day 1 of shorts wear
  A GAITRite system will be used to assess spatio-temporal gait parameters. Participants will walk 4 times over a 5.18m walkway.
Variability of stride width | At baseline and on Day 1 of shorts wear
  A GAITRite system will be used to assess spatio-temporal gait parameters. Participants will walk 4 times over a 5.18m walkway.
Trunk stability in walking | At baseline and on Day 1 of shorts wear
  Acceleration of the trunk and pelvis during gait will be assessed with inertial movement sensors.
Walking speed | At baseline and on Day 1 of shorts wear
  Timed 25-foot walk (T25FW)
Cognitive demand of walking | At baseline and on Day 1 of shorts wear
  Dual task cost will be calculated using the T25FW. Participants will be asked to walk as fast as possible whilst naming alternate letters of the alphabet. The percentage change in walking speed will be calculated, compared to the T25FW assessed without a cognitive task.
Participant rated perception of effect | On Day 1 of shorts wear
  Assessed with a Global Rating of Change scale
Self-perceived walking ability | At baseline and after two weeks of shorts wear
  12-item Multiple Sclerosis Walking Scale
Balance confidence | At baseline and after two weeks of shorts wear
  Activities Specific Balance Confidence scale (ABC),
Frequency of falls | At baseline and after two weeks of shorts wear
  Falls diary

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Following study completion, anonymised data on walking ability with and without orthotic shorts will be made available via the Sheffield Hallam University Research Data Archive.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: All anonymised data will be archived into the Sheffield Hallam University Research Data Archive in September 2019 at which point it will be openly available. This will not include interview recordings or transcripts because of the risk of participants being identied from this data.
Access Criteria: Data will be available as Open Access.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03164031/Prot_SAP_ICF_000.pdf